CLINICAL TRIAL: NCT07272577
Title: Efficacy of Erector Spinae Plane Block on Postoperative Analgesia in Patients Undergoing Laparoscopic Abdominal Surgeries
Brief Title: Erector Spinae Plane Block on Postoperative Analgesia in Patients Undergoing Laparoscopic Abdominal Surgeries
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Bahaa Gamal Saad Mohamed, Anesthesia and Intensive Care, Faculty of Medicine, Assiut University, Assiut, Egypt., Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 618
Record Dates: First submitted 2025-11-27; First posted 2025-12-09 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Erector Spinae Plane Block; Postoperative Analgesia; Laparoscopic Abdominal Surgeries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Erector spinae plane block group (Experimental): Patients will receive an ultrasound-guided erector spinae plane block.
  Interventions: Other: Erector spinae plane block
- Control group (No Intervention): The block will not be performed, and the patients will be shifted to the operation room.

INTERVENTIONS:
Other: Erector spinae plane block — Patients will receive an ultrasound-guided erector spinae plane block.
  Arms: Erector spinae plane block group

SUMMARY:
This study aims to evaluate the efficacy of the erector spinae plane block (ESPB) on postoperative analgesia in patients undergoing laparoscopic abdominal surgeries.

DETAILED DESCRIPTION:
Laparoscopic surgery is associated with less pain, fewer wound infections, reduced hospital stay, reduced morbidity and mortality, and early return to work and improved overall quality of life.

The role of ESPB as a better analgesic modality in reducing 24-hour opioid consumption has recently been established for post-operative analgesia in breast surgeries, video-assisted thoracoscopic surgery, and cardiothoracic surgeries.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Both sexes.
* American Society of Anesthesiologists (ASA) physical status I-II.
* Body mass index (BMI) between 20-30 kg/m2.
* Patients undergoing laparoscopic abdominal surgeries under general anesthesia.

Exclusion Criteria:

* Bleeding or coagulation disorders.
* Having local sepsis, pre-existing.
* Peripheral neuropathies.
* Chronic pain conditions.
* Having any contraindication to regional anesthesia administration.
* Opioid dependency.
* Hypertension.
* Uncontrolled diabetes mellitus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-12-10 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Time to the 1st rescue analgesia | 24 hours postoperatively
  Time to the first request for the rescue analgesia (time from the end of surgery to first dose of morphine administrated).

SECONDARY OUTCOMES:
Total morphine consumption | 24 hours postoperatively
  Rescue analgesia of morphine will be given as 3 mg bolus if the Visual Analogue Scale (VAS) > 3 to be repeated after 30 min if pain persists until the VAS < 4.
Mean arterial pressure | Till the end of surgery (Up to 2 hours)
  Mean arterial pressure will be recorded before skin incision, one minute after skin incision and then recorded regularly every 10 minutes.
Heart rate | Till the end of surgery (Up to 2 hours)
  Heart rate will be recorded before skin incision, one minute after skin incision and then recorded regularly every 10 minutes.
Degree of pain | 24 hours postoperatively
  Each patient will be instructed about postoperative pain assessment with the Visual Analogue Scale (VAS). VAS (0 represents "no pain" while 10 represents "the worst pain imaginable"). VAS will be assessed at 0, 4, 6, 8, 12, and 24 h postoperatively.
Incidence of adverse events | 24 hours postoperatively
  Incidence of adverse events such as bradycardia, hypotension, nausea, vomiting, respiratory depression, or any other complication were recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author